CLINICAL TRIAL: NCT06069609
Title: Orientation Characteristics of Kalifilcon A Daily Disposable Toric Contact Lenses Compared to Acuvue Oasys 1-Day for Astigmatism Contact Lenses
Brief Title: Orientation Characteristics of Daily Disposable Toric Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ROC2-23-006
Record Dates: First submitted 2023-09-19; First posted 2023-10-06 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Astigmatism
Keywords: Contact Lens
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- kalifilcon A Daily Disposable Toric (Experimental)
  Interventions: Device: kalifilcon A Daily Disposable Toric
- Acuvue Oasys 1-Day for Astigmatism (Active Comparator)
  Interventions: Device: Acuvue Oasys 1-Day for Astigmatism

INTERVENTIONS:
Device: kalifilcon A Daily Disposable Toric — kalifilcon A Daily Disposable Toric
  Arms: kalifilcon A Daily Disposable Toric
Device: Acuvue Oasys 1-Day for Astigmatism — Acuvue Oasys 1-Day for Astigmatism
  Arms: Acuvue Oasys 1-Day for Astigmatism

SUMMARY:
Brief summary: Approximately 30 soft toric contact lens adapted subjects will be enrolled in this feasibility, bilateral, randomized, double-masked (subject and investigator), repeated measures insertion study.

DETAILED DESCRIPTION:
Approximately 30 soft toric contact lens adapted subjects will be enrolled in this feasibility, bilateral, randomized, double-masked (subject and investigator), repeated measures insertion study. All subjects will be seen for a Screening/Dispensing Visit at which informed consent will be obtained and eligibility will be assessed. If subjects satisfy all eligibility criteria, subjects will be dispensed study lenses according to unique randomization tables that will be provided to each Investigator. If study eligibility is met, subjects will have lenses inserted in random, successive order. Subjects will be receiving each of the study lens types once, in a randomized order. The subject will wear each of the study contact lenses for approximately 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years or older on the date the Informed Consent Form (ICF) is signed and have capacity to read, understand and provide written voluntary informed consent.
2. Have physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings.
3. Have no active ocular disease or allergic conjunctivitis
4. Not be using any topical ocular medications.
5. Be willing and able to follow instructions.
6. Have signed a statement of informed consent.

Exclusion Criteria:

The subject is not eligible to participate in the study if the subject is:

1. Participating in a conflicting study in the opinion of the Investigator.
2. Considered by the Investigator to not be a suitable candidate for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bausch & Lomb, Incorporated, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 Subjects were screened for eligibility between August 11, 2023 and August 15, 2023.
Pre-assignment Details: 30 of 30 subjects were randomized.
Groups:
- Participants Received Kalifilcon A Daily Disposable Toric and Acuvue Oasys 1-Day for Astigmatism: Participants first received kalifilcon A Daily Disposable Toric then received control lens on day of study visit.
Period: Overall Study
Arm/Group | Participants Received Kalifilcon A Daily Disposable Toric and Acuvue Oasys 1-Day for Astigmatism
Started | 30
Kalifilcon A Daily Disposable Toric | 30
Acuvue Oasys 1-Day for Astigmatism | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants Received Kalifilcon A Daily Disposable Toric and Acuvue Oasys 1-Day for Astigmatism: All 30 subjects that completed the study received both kalifilcon A Daily Disposable Toric and Acuvue Oasys 1-Day for Astigmatism
Arm/Group | Participants Received Kalifilcon A Daily Disposable Toric and Acuvue Oasys 1-Day for Astigmatism
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (12.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race : Asian | 1
  Race : Black or African American | 1
  Race : More than one race | 1
  Race : White | 27
  Ethnicity : Hispanic or Latino | 0
  Ethnicity : Not Hispanic or Latino | 28
  Ethnicity : Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Primary Gaze Orientation
Description: Primary gaze orientation 5 minutes after lens insertion
Time Frame: Assessed 5 minutes after lens insertion
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Participants Received Kalifilcon A Daily Disposable Toric and Acuvue Oasys 1-Day for Astigmatism
Number analyzed (Participants) | 30
Degrees
  kalifilcon A toric lenses at 5 min | 2.4 (3.62)
  Acuvue Oasys 1-Day for Astigmatism at 5 min | 7.9 (13.54)

ADVERSE EVENTS:
Time Frame: Assessed for approximately 30 minutes
Description: There were no adverse events.
Arm/Group | Participants Received Kalifilcon A Daily Disposable Toric and Acuvue Oasys 1-Day for Astigmatism
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/09/NCT06069609/Prot_SAP_001.pdf